CLINICAL TRIAL: NCT05736081
Title: Short-term Effect of Intravitreal Dexamethasone Implant in Refractory Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE-20-13
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema; Ozurdex; Dexamethasone intravitreal implant
MeSH Terms: interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravitreal dexamethasone implant (Experimental): All patients were included here and received one intravitreal dexamethasone implant 0.7mg
  Interventions: Drug: Intravitreal dexamethasone implant

INTERVENTIONS:
Drug: Intravitreal dexamethasone implant — Intravitreal implant of dexamethasone 0.7 mg with previous topic anesthesia and iodine drops
  Other Names: Ozurdex implant

SUMMARY:
The goal of this clinical trial es to learn about the short term effects of intravitreal dexamethasone implant (IDI) in patients with refractory diabetic macular edema. The main question it aims to answer is:

How fast does the diminishing in central retinal thickness has statistical significance after IDI in patients with refractory diabetic macular edema? Patients will be evaluated by OCT before and after the implant.

DETAILED DESCRIPTION:
Patients were evaluated at baseline, 2 hours, 3 hours, 24 hours, 1 week and 1 month post IDI

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 or type 2 diabetes
* diabetic macular edema involving the foveal center with CRT >300 μm measured by OCT
* at least 3 and maximum 9 monthly intravitreal injections of anti-VEGF

Exclusion Criteria:

* uncontrolled diabetes (blood glucose ≥ 250 mg/dL at any time
* previous IDI
* any condition precluding adequate fundus visualization
* uncontrolled glaucoma
* papillary excavation ≥ 0.7

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in central retinal thickness | Prospective: from baseline to 2 hours, 3 hours, 24 hours, 1 week and 1 month post IDI
  Difference among the baseline and the posterior measurements of the CRT with OCT

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity | Prospective: from baseline to 1 month post IDI
  Measurement of Best Corrected Visual Acuity before and after IDI

CONTACTS AND LOCATIONS:
Overall Officials: José Gerardo García Aguirre, MD, Principal Investigator — Asociación para Evitar la Ceguera en México I.A.P.
Locations (1):
- Asociacion Para Evitar la Ceguera en Mexico, Mexico City, Coyoacan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available when the summary date are published
Access Criteria: VIa e-mail with José Gerardo García Aguirre MD, all IPD that underlie results in a publication will be available

REFERENCES:
- [Background] Tang J, Kern TS. Inflammation in diabetic retinopathy. Prog Retin Eye Res. 2011 Sep;30(5):343-58. doi: 10.1016/j.preteyeres.2011.05.002. Epub 2011 May 25. PMID 21635964
- [Background] Noma H, Yasuda K, Shimura M. Involvement of Cytokines in the Pathogenesis of Diabetic Macular Edema. Int J Mol Sci. 2021 Mar 26;22(7):3427. doi: 10.3390/ijms22073427. PMID 33810434
- [Background] Wallsh JO, Gallemore RP. Anti-VEGF-Resistant Retinal Diseases: A Review of the Latest Treatment Options. Cells. 2021 Apr 29;10(5):1049. doi: 10.3390/cells10051049. PMID 33946803
- [Background] Bressler SB, Ayala AR, Bressler NM, Melia M, Qin H, Ferris FL 3rd, Flaxel CJ, Friedman SM, Glassman AR, Jampol LM, Rauser ME; Diabetic Retinopathy Clinical Research Network. Persistent Macular Thickening After Ranibizumab Treatment for Diabetic Macular Edema With Vision Impairment. JAMA Ophthalmol. 2016 Mar;134(3):278-85. doi: 10.1001/jamaophthalmol.2015.5346. PMID 26746868
- [Background] Boyer DS, Yoon YH, Belfort R Jr, Bandello F, Maturi RK, Augustin AJ, Li XY, Cui H, Hashad Y, Whitcup SM; Ozurdex MEAD Study Group. Three-year, randomized, sham-controlled trial of dexamethasone intravitreal implant in patients with diabetic macular edema. Ophthalmology. 2014 Oct;121(10):1904-14. doi: 10.1016/j.ophtha.2014.04.024. Epub 2014 Jun 4. PMID 24907062
- [Background] Khan Z, Kuriakose RK, Khan M, Chin EK, Almeida DR. Efficacy of the Intravitreal Sustained-Release Dexamethasone Implant for Diabetic Macular Edema Refractory to Anti-Vascular Endothelial Growth Factor Therapy: Meta-Analysis and Clinical Implications. Ophthalmic Surg Lasers Imaging Retina. 2017 Feb 1;48(2):160-166. doi: 10.3928/23258160-20170130-10. PMID 28195619
- [Derived] Moreno JB, Medina DB, Rosellon-Escobar MF, Garcia-Aguirre JG. Short-term effect of intravitreal dexamethasone implant in refractory diabetic macular edema. BMC Ophthalmol. 2024 Mar 11;24(1):113. doi: 10.1186/s12886-024-03341-9. PMID 38462613